## FRUIT-MAIC

| Version | 1.0 |
|---|---|
| Date | 1 <sup>st</sup> August 2025 |
| Brief Title | Match-Adjusted Indirect Comparison (MAIC) of Fruquintinib plus Paclitaxel versus Ramucirumab |
| | plus Paclitaxel in Advanced Gastric/GEJ Adenocarcinoma |
| Acronym | FRUIT-MAIC |
| Sponsor | |
| Information provided by | |
| Brief Summary | This anchored matching-adjusted indirect comparison (MAIC) evaluates the relative efficacy of |
| | fruquintinib-paclitaxel (using IPD from the FRUTIGA trial, n=703) versus ramucirumab-paclitaxel |
| | (using published AgD from RAINBOW-Asia, n=440) in advanced gastric/GEJ adenocarcinoma. |
| | Baseline characteristics are adjusted via entropy balancing weights. Primary endpoint is progression- |
| | free survival (PFS) analyzed by Bucher method; secondary endpoints include overall survival (OS) |
| | and objective response rate (ORR). Sensitivity analyses comprise restricted mean survival time |
| | (RMST) analysis and simulated treatment comparison (STC). |
| Detailed Description | This retrospective MAIC analysis employs individual patient data (IPD) from the FRUTIGA trial |
| | (fruquintinib arm) and published aggregate data (AgD) from RAINBOW-Asia (ramucirumab arm), |
| | with placebo as the common anchor. Pseudo individual participant data (Pseudo-IPD) for the |
| | RAINBOW-Asia trial were reconstructed from published Kaplan-Meier curves using the Guyot |
| | algorithm (2012). |
| | Weighting Methodology: |
| | <ul> <li>Seven prognostic factors balanced: age &lt;65, male sex, ECOG 0, GEJ primary, peritoneal<br/>metastases, metastatic sites, prior doublet chemotherapy</li> </ul> |
| | Optimization via BFGS algorithm (convergence tolerance 1e-6) |
| | <ul> <li>Effective sample size (ESS) retention: &gt; 50%</li> </ul> |
| | Statistical Analysis: |
| | <ul> <li>Primary: Adjusted PFS hazard ratio (HR) using Bucher method with 95% bootstrap CI (100 iterations)</li> </ul> |
| | <ul> <li>Secondary: Weighted Cox models for OS; logistic regression for ORR/DCR</li> <li>Sensitivity: Simulated Treatment Comparison (STC) and covariate threshold analyses</li> </ul> |
| | Sensitivity Analyses: |
| | o RMST analyses were conducted as supportive evidence alongside primary Cox models for |
| | time-to-event endpoints violating proportional hazards assumptions. |
| | o Restricted mean survival time (RMST) |
| | o Simulated Treatment Comparison (STC) |
| | Bootstrap confidence intervals (100 iterations) |
| Official Title | Adjusted Indirect Treatment Comparison of Fruquintinib-based Therapy Versus Standard Care in |
| - 44.4 | Advanced Gastric/Gastroesophageal Junction Adenocarcinoma: A MAIC Analysis. |
| Conditions | Advanced Gastric Cancer |
| | Gastroesophageal Junction Adenocarcinoma |
| Intervention/Treatment | Experimental: Fruquintinib + paclitaxel, Ramucirumab + paclitaxel |
| | Common comparator: Placebo + paclitaxel (weighted FRUTIGA and RAINBOW-Asia reference arm) |
| Inclusion Criteria | 1. Histologically confirmed gastric/GEJ adenocarcinoma |
| | 2. Advanced or metastatic disease |
| | 3. ECOG 0-1 |
| | 4. Received either fruquintinib + paclitaxel or reference regimen |
| Evaluation Criteri | 5. Available baseline characteristics for matching variables |
| Exclusion Criteria | 1. Missing key outcome data |
| | 2. Incomplete baseline characteristics for >2 matching variables |
| | 3. Prior fruquintinib exposure (control arm only) |

| Primary Purpose | Treatment Comparison |
|------------------------|--------------------------------------------------|
| Allocation | Observational |
| Interventional Model | Indirect Treatment Comparison |
| Masking | |
| Participant Group/Arm | Group 1: Fruquintinib + Paclitaxel (IPD) |
| | Group 2: Control Therapy (AgD from RAINBOW-Asia) |
| Intervention/Treatment | |

| Primary Outcome Measures | | |
|---|---|---|
| Outcome Measure | Measure Description | Time Frame |
| Progression-Free Survival | Time from randomization to progression/death, | per FRUTIGA trial data cutoff |
| (PFS) | assessed via weighted Cox model | |

| Second Outcome Measures | | |
|---|---|---|
| Outcome Measure | Measure Description | Time Frame |
| Objective Response Rate | CR+PR per RECIST 1.1, compared via weighted | per FRUTIGA trial data cutoff |
| (ORR) | logistic regression | |
| Disease Control Rate | CR+PR+SD≥6 weeks, analyzed via weighted | per FRUTIGA trial data cutoff |
| (DCR) | proportions | |
| Overall Survival (OS) | Time from randomization to death, analyzed using | per FRUTIGA trial data cutoff |
| | weighted Kaplan-Meier | |
| Subgroup Analyses | PFS/OS by ECOG, metastasis burden, primary site, | A |
| | etc. | As per primary outcomes |

| Other Outcome Measures | | |
|---|---|---|
| Outcome Measure | Measure Description | Time Frame |
| Progression-Free Survival | Simulated Treatment Comparison (STC), Bootstrap | per FRUTIGA trial data cutoff |
| (PFS) | confidence intervals (100 iterations) | |